CLINICAL TRIAL: NCT03306342
Title: Clinical Study to Investigate Visual Performance, Patient Satisfaction and PCO Rate After Implantation of a Trifocal Hydrophobic IOL
Brief Title: Visual Performance, Patient Satisfaction and PCO Rate After Implantation of a Trifocal Hydrophobic IOL
Acronym: PHY1703
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY 1703
Record Dates: First submitted 2017-09-27; First posted 2017-10-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Cataract; Lens Opacities; Presbyopia
Keywords: Intraocular Lens; trifocal; hydrophobic; hydrophilic
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IOL implantation experimental (Experimental): hydrophobic, trifocal intraocular lens POD F GF
  Interventions: Device: IOL implantation experimental

INTERVENTIONS:
Device: IOL implantation experimental — Implantation of trifocal IOL POD F GF consisting of hydrophobic material

SUMMARY:
Prospective, controlled, single-surgeon, single-center post-market clinical follow up study to investigate the clinical outcomes of a hydrophobic trifocal IOL (PhysIOL POD F GF)

DETAILED DESCRIPTION:
This clinical investigation is a prospective, controlled, single-surgeon, single-center post-market clinical follow up study whereby patients undergoing routine cataract surgery will have bilateral implantation of trifocal intraocular lenses FineVision POD F GF (PhysIOL, Liège, Belgium).

The study purpose is to obtain clinical data on visual acuity, contrast sensitivity, questionnaire outcomes and PCO rate on patients implanted with FineVision POD F GF.

The device under investigation (FineVision POD F GF) is a trifocal glistening-free hydrophobic acrylic intraocular lens (IOL) manufactured by the sponsor of this study PhysIOL sa/nv. The IOL will be implanted as part of the routine cataract surgery on patients suffering from cataract development.

In total 25 patients will be recruited for this clinical study and receive a bilateral implantation of FineVision POD F GF intraocular lens.

Subjects participating in the trial will attend a total of 8 study visits (1 preoperative, 2 operative and 5 postoperative) over a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Cataractous eyes with no comorbidity
* Spontaneously emitting the desire for spectacle independence after surgery and with realistic expectation.
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent

Exclusion Criteria:

* Irregular astigmatism
* Age of patient < 45 years
* Regular corneal astigmatism >0.75 dioptres by an automatic keratometer or biometer or >1.0 dioptres if the steep axis of cylinder is between 90° and 120° in one or both eyes
* Difficulty for cooperation (distance from their home, general health condition)
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma etc…)
* Any ocular comorbidity
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)
* AMD suspicious eyes (determined by OCT)
* Complicated surgery

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
binocular Uncorrected Distance Visual Acuity (UDVA) | 3 months postoperative
  Statistically significant equality between literature data and data obtained in this study on binocular UDVA. UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014

SECONDARY OUTCOMES:
Manifested refraction | 3 months postoperative
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2014. This data will also be used to calculate the manifested refractive spherical equivalent (MRSE)
Uncorrected Distance Visual Acuity (UDVA) | 3 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Corrected Distance Visual Acuity (CDVA) | 3 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Distance Corrected Intermediate Visual Acuity (DCIVA) | 3 months postoperative
  DCIVA is measured with ETDRS charts placed in 70cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Uncorrected Intermediate Visual Acuity (UIVA) | 3 months postoperative
  UIVA is measured with ETDRS charts placed in 70cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Distance Corrected Near Visual Acuity (DCNVA) | 3 months postoperative
  DCNVA is measured with ETDRS charts placed in 35cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Uncorrected Near Visual Acuity (UNVA) | 3 months postoperative
  UNVA is measured with ETDRS charts placed in 35cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Contrast Sensitivity | 3 months postoperative
  Contrast Sensitivity under photopic and mesopic light conditions using the standardized contrast sensitivity device CSV-1000 (VectorVision)
Aberrometry | 3 months postoperative
  Aberrometry outcomes are measured with a standard aberrometer. The following values will be evaluated in this study: Spherical aberrations, high order aberrations, lens tilt.
PCO rate | 2 years postoperative
  The rate of patients showing posterior capsular opacities (PCO) long term after surgery will be assessed. The criteria is, if the eye requires a secondary treatment to remove the PCO.
questionnaire | 3 months postoperative
  Outcomes measures of a questionnaire to address the general patient satisfaction and possible side effects of the treatment. For this study, the validated and verified questionnaire VFQ-25 (National Eye Institute) will be used. The maximum score for each question is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice Cochener, Prof., Principal Investigator — Département d'ophtalmologie - CHU Morvan Bâtiment 4 bis
Locations (1):
- Département d'ophtalmologie - CHU Morvan Bâtiment 4 bis, Brest, France

IPD SHARING:
Plan to Share IPD: No